CLINICAL TRIAL: NCT02672657
Title: Assessing the Evolution and Determinants of Quality of Life in Elderly Cancer Patients and Their Caregivers: a Prospective Multicenter Observational Cohort Study.
Brief Title: Determinants of Quality Of Life in AGEd Cancer Patients
Acronym: DEQOLAGE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Paris 12 Val de Marne University (Other); Research Team APEMAC EA4360, University of Lorraine (Unknown); Unité de Recherche Clinique Mondor, Hôpital Henri Mondor (Unknown); Institut de Cancérologie de Lorraine (Other); Unité de Coordination en Onco-Gériatrie (UCOG) Sud Val-de-Marne (Unknown); Quality of life and cancer clinical research platform (Unknown); Ligue contre le cancer, France (Other); Conseil Régional de Lorraine, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2014-A00317-40
Record Dates: First submitted 2016-01-14; First posted 2016-02-03 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Colorectal Neoplasms; Prostatic Neoplasms
Keywords: Health-Related Quality of life; Cancer; Elderly; Caregivers
MeSH Terms: conditions — Colorectal Neoplasms; Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients face multiple stresses and challenges in the aftermath of cancer diagnosis. Despite needs perceived by elderly patients might differ from those of younger patients, there is a paucity of published data assessing the specific evolution and relevant determinants of health-related quality of life (HRQoL) in older patients with cancer. Such determinants may include cancer type/location/stage, treatment type/intensity, comorbidities, nutritional status or socioeconomic features, but also practical organization of care -frequency, geographical distance, supporting measures -, or psychosocial and material support - social network, housing conditions and contextual neighborhood features. Comparatively to dementia or cancer in younger patients, little is known in the oncogeriatric field of the impact on caregivers' perceived burden and HRQol of the support they provide to patients. Further, the potential interactions between patients' and caregivers' HRQoL remain largely unknown, while caregivers are often themselves old with chronic diseases and/or daily living activities' limitations.

The DEQOLAGE study is a prospective observational cohort study that aims to describe the HRQoL of patients aged over 70 years with a colorectal or prostatic cancer during the first year following the diagnosis of the disease as well as the HRQoL and burden in their main caregivers. This study will allow a comprehensive assessment of multiple determinants of HRQoL operating at different levels, including individual (cancer type/location/stage, treatment type/intensity, comorbidities, nutritional status or socioeconomic features), contextual (social network, housing conditions and contextual neighborhood features) and organizational factors (frequency, geographical distance, supporting measures). We also hypothesize that complex interactions may operate between patient's and caregiver's HRQoL and perceived burden. Quality of life measurement will be based on two recent scales specifically designed for the elderly to confirm their psychometric properties and in-field feasibility.

ELIGIBILITY:
Patients

Inclusion Criteria:

* Aged 70 or more
* With a new histologically confirmed diagnosis of colorectal or prostate cancer
* With a Comprehensive Geriatric Assessment (CGA) performed before the initiation of cancer treatment
* Having expressed their oral non-opposition to participate in the study
* Affiliated to a health insurance scheme

Exclusion Criteria:

* Expected survival inferior to 6 months, based on the clinical appreciation from the physician in charge of the enrollment
* Cancer recurrence in patients previously treated
* Physical, cognitive or linguistic incapacity to complete questionnaires

Caregivers Inclusion criteria

* Aged 18 or more
* Nonprofessionally, partially or fully helping the patient in daily activities and accompanying the patient to visits; familial ties with the patient are not required (spouse, child, friend or neighbor)
* In contact with the patient more than once a week
* Defined by the patient during the inclusion visit as the main caregiver

Exclusion criteria

- Physical, cognitive or linguistic incapacity to complete questionnaires

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients presenting at the participating hospitals with newly diagnosed colorectal or prostate cancer and referred by an oncologist, surgeon, radiotherapist, or other specialist to the hospital geriatric oncology clinics for a multidimensional geriatric assessment before the initiation of cancer treatment will be eligible for inclusion, regardless of stage at diagnosis and plans for treatment
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-02; Primary Completion 2019-02 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Changes in HRQoL of patients and their caregivers as assessed by the generic WHOQOL-BREF questionnaires | At baseline, 3, 6, and 12 months
Changes in HRQoL of patients and their caregivers if aged >70 years as assessed by the WHOQOL-OLD questionnaire | At baseline, 3, 6, and 12 months
Changes in HRQoL of patients as assessed by the specific EORTC-QLQ C30 questionnaire | At baseline, 3, 6, and 12 months
Changes in HRQoL of patients as assessed by the specific EORTC QLQ-ELD14 questionnaire | At baseline, 3, 6, and 12 months
Changes in burden of patients' caregivers as assessed by the Zarit burden inventory questionnaire | At baseline, 3, 6, and 12 months

SECONDARY OUTCOMES:
Psychometric properties of the HRQoL questionnaire WHOQOL-OLD (validity, reliability, sensitivity to change, feasibility) | At baseline, 3, 6, and 12 months
Psychometric properties of the HRQoL questionnaire EORTC QLQ-ELD14 (validity, reliability, sensitivity to change, feasibility) | At baseline, 3, 6, and 12 months
Prognostic value of baseline HRQoL measurements on cancer progression-free survival | At baseline, 3, 6, and 12 months
Prognostic value of baseline HRQoL measurements on overall survival | At baseline, 3, 6, and 12 months
Prognostic value of baseline HRQoL measurements on patient's functional decline, defined as any decrease in the ADL scale | At baseline, 3, 6, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Christine Perret-Guillaume, Study Chair — Central Hospital, Nancy, France; Elena Paillaud, Study Chair — Hôpital Albert Chenevier
Locations (3):
- France (3):
  - Hôpital Henri Mondor, Créteil
  - CHRU Nancy, Nancy
  - Hôpital Saint Louis, Paris

IPD SHARING:
Plan to Share IPD: No